CLINICAL TRIAL: NCT04551482
Title: Oxytocin as a Neuroendocrine Therapy for Obesity in Youth
Brief Title: Oxytocin for Weight Loss in Adolescents
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Elizabeth Austen Lawson, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020P002511; 1R01DK124223-01A1 (NIH)
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Obesity, Adolescent; Oxytocin
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Experimental): Oxytocin nasal spray (24 IU nasal spray, 4 times per day for 12 weeks)
  Interventions: Drug: Oxytocin nasal spray
- Placebo (Placebo Comparator): Placebo nasal spray (24 IU nasal spray, 4 times per day for 12 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — 24 IU nasal spray, 4 times per day for 12 weeks
  Other Names: Syntocin
  Arms: Oxytocin
Drug: Placebo — 24 IU nasal spray, 4 times per day for 12 weeks
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo-controlled study of the effects of intranasal oxytocin in youths with obesity, ages 12-18 years old. Subjects will be randomized to receive intranasal oxytocin or placebo (1 spray per nostril, 4 times per day) for 12 weeks. Study visits include screening to determine eligibility, 2-part main study visits at baseline, week 8, and week 12, and safety check-in visits at weeks 1, and 4; phone calls at weeks 2, 6, and 10, with a safety follow-up visit 6 weeks after the last dose of study drug. Study procedures include appetite, behavioral, metabolic, and endocrine assessments.

DETAILED DESCRIPTION:
In recent years there has been a dramatic increase in obesity and its complications in both children and adults. Earlier treatment substantially reduces the likelihood of developing complications later in life while concurrently improving quality of life and decreasing mortality. Therefore, it is essential to develop safe and effective therapeutic strategies for weight loss, particularly in adolescents. Oxytocin (OXT), a hypothalamic peptide hormone that regulates energy balance, is a novel neuroendocrine weight-loss therapeutic in adults with obesity because it simultaneously reduces energy intake and increases energy expenditure and is well-tolerated. Data are currently lacking regarding effects of OXT administration in adolescents with obesity.

The current study is a 12-week randomized controlled trial (RCT) of OXT vs. placebo in 12-18-year old adolescents with obesity. We hypothesize that OXT administration will decrease weight as a consequence of decreased caloric intake and increased energy expenditure, both partially mediated by reduced hypothalamic inflammation (such inflammation drives weight gain by increasing food intake and reducing energy expenditure). Further, OXT will improve metabolic risk markers, such as visceral and intrahepatic fat, systemic inflammation, and serum lipids.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, 10-18 years
* Obesity (BMI ≥95th percentile for age and gender)
* Willingness to maintain current diet and lifestyle for the duration of study participation

Exclusion Criteria:

* Active substance abuse
* Use of prescription or over-the-counter drugs or dietary/herbal supplements for the purpose of weight loss. Medications/supplements that may affect weight will be allowed if participants are on a stable dose with stable weight for at least 3 months.
* Greater than 5kg weight loss over 3 months;
* Follows a nonstandard diet (e.g., gluten-free, vegan, Paleo, Atkins, raw diet, macrobiotic diet)
* Cardiovascular disease
* Prolonged QT interval
* Chronic gastrointestinal disorders and other inflammatory conditions
* Epilepsy
* Untreated thyroid disease
* Alanine transaminase (ALT) or aspartate transaminase (AST) >2.5 times upper limit of normal
* Creatinine >1.5 mg/dl
* Hyponatremia
* Pregnancy/breastfeeding or refusal to use contraception not containing estrogen throughout the study if female and sexually active
* MRI exclusion criteria such as the presence of a pacemaker or cerebral aneurysm clips
* Weight >450 lbs due to limits for MRI and DXA scanners
* Type 1 Diabetes Mellitus or Type 2 Diabetes Mellitus if HbA1c >8%
* Active eating disorder

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Weight | 12 weeks
  Mean difference in weight between Oxytocin and Placebo group after 12 weeks of treatment
Height | Baseline
  Measure height on a stadiometer to the nearest 0.1 cm
Body mass index (BMI) | 12 weeks
  Mean difference in BMI between Oxytocin and Placebo group after 12 weeks of treatment. BMI will be calculated as weight/height2

SECONDARY OUTCOMES:
Lean mass and Fat mass | 12 weeks
  Dual Energy Absorptiometry (DXA) will be used for measuring fat mass (kg) and lean mass (Kg)
Fasting Resting Energy Expenditure (kCal) | 12 weeks
  Assessed by Indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lawson, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No